CLINICAL TRIAL: NCT04464187
Title: Prospective Registry to Evaluate Pregnancy Outcomes in Women Treated With Elagolix
Brief Title: A Study to Evaluate Pregnancy Outcomes in Females Treated With Oral Elagolix Tablets and Capsules
Status: Terminated | Type: Observational
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P18-954
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Uterine Fibrioids
Keywords: Endometriosis; Pregnancy; Orlissa; Elagolix; Uterine fibriods; Oriahnn
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants exposed to Elagolix-containing products: Pregnant participants exposed to Elagolix from 14 days after last menstrual period (LMP) or at any point during pregnancy.
- Participants not exposed to Elagolix-containing products: Pregnant participants with endometriosis, uterine fibroids, or other conditions based on approved indications and prescribing patterns of Elagolix-containing products not exposed to Elagolix from 14 days after LMP or at any point during pregnancy.

SUMMARY:
Orilissa is a drug approved for the management of moderate to severe pain associated with endometriosis. Oriahnn is approved for heavy menstrual bleeding due to uterine fibroids. Elagolix-containing products should not be taken by women who are pregnant or suspected to be pregnant but pregnancies are expected as the medicine does not completely stop ovulation and women may inadvertently continue taking Elagolix-containing products until their pregnancy is confirmed.

This study will assess pregnancy outcomes (maternal, fetal, and infant) of participants with and without exposure to Elagolix-containing products for their endometriosis or other conditions based on approved indications and prescribing patterns of Elagolix. Around 584 participants will be enrolled (292 participants exposed to Elagolix and 292 without exposure) in the United States.

Participants will not receive Elagolix-containing products as part of this study but will be followed for maternal and fetal outcomes up to 1 year after delivery.

There may be a higher burden for participants in this study compared to standard of care. Participants will be asked to provide additional information by questionnaire during each trimester of pregnancy, and at 0-6 weeks, 26 weeks, and 1 year after delivery. Contact Bloom Pregnancy Call Center at 1-833-782-7241 or bloompregnancyregistry@iqvia.com or visit https://www.bloompregnancyregistry.com/.

ELIGIBILITY:
Inclusion Criteria:

Participants exposed to Elagolix:

* Currently pregnant.
* Documentation that the participant was exposed to elagolix-containing product from 14 days after last menstrual period (LMP) or at any time during pregnancy.
* Consents to participate in the study. If the participant is a minor, consent will be obtained according to local regulations.

Internal Comparator:

* Currently pregnant with endometriosis, uterine fibroids, or other conditions based on approved indications and prescribing patterns of elagolix-containing product.
* Documentation that the participant was not exposed to elagolix-containing product from 14 days after LMP or any time during pregnancy.
* Consents to participate in the study. If the participant is a minor, consent will be obtained according to local regulations.

Exclusion Criteria:

-None.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with or without exposure to Orilissa for their endometriosis or other indications for prescribing of the medication.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Rate of major congenital malformations | Approximately 2 years (1 year post-delivery)
  Defined as an abnormality in structural development that is medically or cosmetically significant, present at birth, and persists in postnatal life unless or until repaired.

SECONDARY OUTCOMES:
Rate of minor congenital malformations | Approximately 2 years (1 year post-delivery)
  Defined as a defect that occurs infrequently in the population but that has neither cosmetic nor functional significance to the child and is identified in the infant up to 1 year of age.
Rate of spontaneous abortion | Up to 9 months
  Defined as non-deliberate embryonic or fetal death that occurs prior to 20 weeks gestation post-last menstrual period.
Rate of elective or therapeutic pregnancy termination | Up to 9 months
  Rate of elective or therapeutic pregnancy termination.
Rate of stillbirth | Up to 9 months
  Defined as non-deliberate fetal death that occurs at or after 20 weeks gestation but prior to delivery.
Rate of preterm birth | Up to 9 months
  Defined as live birth prior to 37 weeks gestation as counted from last menstrual period or based on ultrasound used for conception dating.
Rate of maternal placental issues | Up to 9 months
  Rate of maternal placental issues, including placenta previa and placental abruption.
Rate of small for gestation age infants | Up to 9 months
  Defined as birth size (weight, length, or head circumference) less than or equal to the 10th percentile for sex and gestational age using National Center for Health Statistics (NCHS) pediatric growth curves for full-term infants. Prenatal growth curves specific to preterm infants will be used for premature infants.
Rate of postnatal growth deficiency or failure to thrive | Approximately 2 years (1 year post-delivery)
  Rate of postnatal growth deficiency or failure to thrive as diagnosed by his/her treating physician using criteria such as a significant weight or weight-for-height deceleration.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Iqvia /Id# 240918, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info. — https://www.bloompregnancyregistry.com/